CLINICAL TRIAL: NCT07324434
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 1 Study of Oral F-02-2-Na Tablets in Adult Subjects: Assessment of the Safety and Pharmacokinetics of Single Ascending Doses (to Include the Mass Balance) & Multiple Ascending Doses
Brief Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Oral F-02-2-Na Tablets in Adult Subjects
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Hengqin Novagains Biopharmaceutical Co., Ltd. (Industry)
Collaborators: Xiangbei Welman Pharmaceutical Co., Ltd (Industry); Guangzhou Xin-Chuangyi Biopharmaceutical Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F-02-2-Na-2025-PROT-I-1
Record Dates: First submitted 2025-11-28; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Hyperuricemia With or Without Gout

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (18):
- A1-0.5mg T (Experimental): The intervention consists of a single oral administration of F-02-2-Na (0.5 mg). The study drug is administered in a fasting state (at least 10 hours), and subjects will be continuously monitored for 72 hours following administration in Safety and PKPD assessments.
  Interventions: Drug: F-02-2-Na Tablet (0.5 mg)
- A1-0.5mg R (Placebo Comparator): The intervention consists of a single oral administration of matching placebo (0.5mg). The administration conditions are the same as those for the experimental arm
  Interventions: Drug: F-02-2-Na Matching Placebo (0.5mg)
- A2-5mg-T (Experimental): The intervention consists of a single oral administration of F-02-2-Na (5 mg). The study drug is administered in a fasting state (at least 10 hours), and subjects will be continuously monitored for 72 hours following administration in Safety and PKPD assessments
  Interventions: Drug: F-02-2-Na Tablet (5mg)
- A2-5mg-R (Placebo Comparator): The intervention consists of a single oral administration of matching placebo (5mg). The administration conditions are the same as those for the experimental arm.
  Interventions: Drug: F-02-2-Na Matching Placebo (5mg)
- A3-25mg-T (Experimental): The intervention consists of a single oral administration of F-02-2-Na (25 mg). The study drug is administered in a fasting state (at least 10 hours), and subjects will be continuously monitored for 72 hours following administration in Safety and PKPD assessments.
  Interventions: Drug: F-02-2-Na Tablet (25mg)
- A3-25mg-R (Placebo Comparator): The intervention consists of a single oral administration of matching placebo (25mg). The administration conditions are the same as those for the experimental arm.
  Interventions: Drug: F-02-2-Na Matching Placebo (25mg)
- A4-75mg-T (Experimental): The intervention consists of a single oral administration of F-02-2-Na (75 mg). The study drug is administered in a fasting state (at least 10 hours), and subjects will be continuously monitored for 72 hours following administration in Safety and PKPD assessments.
  Interventions: Drug: F-02-2-Na Tablet (75mg)
- A4-75mg-R (Placebo Comparator): The intervention consists of a single oral administration of matching placebo (75mg). The administration conditions are the same as those for the experimental arm.
  Interventions: Drug: F-02-2-Na Matching Placebo (75mg)
- A5-150mg-T (Experimental): The intervention consists of a single oral administration of F-02-2-Na (150 mg). The study drug is administered in a fasting state (at least 10 hours), and subjects will be continuously monitored for 72 hours following administration in Safety and PKPD assessments
  Interventions: Drug: F-02-2-Na Tablet (150 mg)
- A5-150mg-R (Placebo Comparator): The intervention consists of a single oral administration of matching placebo (150mg). The administration conditions are the same as those for the experimental arm.
  Interventions: Drug: F-02-2-Na Matching Placebo (150 mg)
- A6-200mg-T (Experimental): The intervention consists of a single oral administration of F-02-2-Na (200 mg). The study drug is administered in a fasting state (at least 10 hours), and subjects will be continuously monitored for 72 hours following administration in Safety and PKPD assessments.
  Interventions: Drug: F-02-2-Na Tablet (200 mg)
- A6-200mg-R (Placebo Comparator): The intervention consists of a single oral administration of matching placebo (200mg). The administration conditions are the same as those for the experimental arm.
  Interventions: Drug: F-02-2-Na Matching Placebo (200 mg)
- B1-25mg-T (Experimental): The intervention consists of the multiple oral administrations of F-02-2-Na tablets at a dose of 25mg for 7 consecutive days.
  Interventions: Drug: F-02-2-Na Tablet (25mg)-Multiple dose
- B1-25mg-R (Placebo Comparator): The intervention consists of the multiple oral administrations of matching placebo (25mg). The administration conditions are the same as those for the experimental arm.
  Interventions: Drug: F-02-2-Na Matching Placebo (25mg) -Multiple dose
- B2-50mg-T (Experimental): The intervention consists of the multiple oral administrations of F-02-2-Na tablets at a dose of 50mg for 7 consecutive days.
  Interventions: Drug: F-02-2-Na Tablet (50mg)-Multiple dose
- B2-50mg-R (Placebo Comparator): The intervention consists of the multiple oral administrations of matching placebo (50mg). The administration conditions are the same as those for the experimental arm.
  Interventions: Drug: F-02-2-Na Matching Placebo (50mg) -Multiple dose
- B3-100mg-T (Experimental): The intervention consists of the multiple oral administrations of F-02-2-Na tablets at a dose of 100mg for 7 consecutive days.
  Interventions: Drug: F-02-2-Na Matching Placebo (100mg) -Multiple dose
- B3-100mg-R (Placebo Comparator): The intervention consists of the multiple oral administrations of matching placebo (100mg). The administration conditions are the same as those for the experimental arm.
  Interventions: Drug: F-02-2-Na Tablet (100mg)-Multiple dose

INTERVENTIONS:
Drug: F-02-2-Na Tablet (0.5 mg) — The intervention involves the single oral administration of F-02-2-Na tablets at a dose of 0.5 mg, given once in a fasting state (after at least 10 hours of fasting). The drug is formulated as film-coated tablets with a strength of 1 mg per tablet, manufactured by Guangdong Hengqin Novagains Biopharmaceutical Co., Ltd. (batch number: 250901). Safety and PKPD parameters will be continuously monitored for 72 hours following administration.
  Other Names: A1-0.5mg T
  Arms: A1-0.5mg T
Drug: F-02-2-Na Matching Placebo (0.5mg) — The intervention consists of the single oral administration of a matching placebo (0.5mg) for F-02-2-Na. Formulated as film-coated tablets (consistent with F-02-2-Na in appearance, color, and strength), the placebo contains no F-02-2-Na or other pharmacologically active ingredients and is manufactured by Guangdong Hengqin Novagains Biopharmaceutical Co., Ltd. (batch number: 250101). The administration conditions are identical to those of the experimental arm in this study; however, it has no therapeutic effect.
  Other Names: A1-0.5mg R
  Arms: A1-0.5mg R
Drug: F-02-2-Na Tablet (5mg) — The intervention involves the single oral administration of F-02-2-Na tablets at a dose of 5mg, given once in a fasting state (after at least 10 hours of fasting). The drug is formulated as film-coated tablets with a strength of 5mg per tablet, manufactured by Guangdong Hengqin Novagains Biopharmaceutical Co., Ltd. (batch number: 250101). Safety and PKPD parameters will be continuously monitored for 72 hours following administration.
  Other Names: A2-5mg-T
  Arms: A2-5mg-T
Drug: F-02-2-Na Matching Placebo (5mg) — The intervention consists of the single oral administration of a matching placebo (5mg) for F-02-2-Na. Formulated as film-coated tablets (consistent with F-02-2-Na in appearance, color, and strength), the placebo contains no F-02-2-Na or other pharmacologically active ingredients and is manufactured by Guangdong Hengqin Novagains Biopharmaceutical Co., Ltd. (batch number: 250101). The administration conditions are identical to those of the experimental arm in this study; however, it has no therapeutic effect.
  Other Names: A2-5mg-R
  Arms: A2-5mg-R
Drug: F-02-2-Na Tablet (25mg) — The intervention involves the single oral administration of F-02-2-Na tablets at a dose of 25mg, given once in a fasting state (after at least 10 hours of fasting). The drug is formulated as film-coated tablets with a strength of 5mg/10mg per tablet, manufactured by Guangdong Hengqin Novagains Biopharmaceutical Co., Ltd. (batch number: 250101). Safety and PKPD parameters will be continuously monitored for 72 hours following administration.
  In SAD A3 (25 mg), collected blood, urine, and feces will be used for the mass balance study.
  Other Names: A3-25mg-T
  Arms: A3-25mg-T
Drug: F-02-2-Na Matching Placebo (25mg) — The intervention consists of the single oral administration of a matching placebo (25mg) for F-02-2-Na. Formulated as film-coated tablets (consistent with F-02-2-Na in appearance, color, and strength), the placebo contains no F-02-2-Na or other pharmacologically active ingredients and is manufactured by Guangdong Hengqin Novagains Biopharmaceutical Co., Ltd. (batch number: 250101). The administration conditions are identical to those of the experimental arm in this study; however, it has no therapeutic effect.
  Other Names: A3-25mg-R
  Arms: A3-25mg-R
Drug: F-02-2-Na Tablet (75mg) — The intervention involves the single oral administration of F-02-2-Na tablets at a dose of 75mg, given once in a fasting state (after at least 10 hours of fasting). The drug is formulated as film-coated tablets with a strength of 5mg/10mg/50mg per tablet, manufactured by Guangdong Hengqin Novagains Biopharmaceutical Co., Ltd. (batch number: 250101). Safety and PKPD parameters will be continuously monitored for 72 hours following administration.
  Other Names: A4-75mg-T
  Arms: A4-75mg-T
Drug: F-02-2-Na Matching Placebo (75mg) — The intervention consists of the single oral administration of a matching placebo (75mg) for F-02-2-Na. Formulated as film-coated tablets (consistent with F-02-2-Na in appearance, color, and strength), the placebo contains no F-02-2-Na or other pharmacologically active ingredients and is manufactured by Guangdong Hengqin Novagains Biopharmaceutical Co., Ltd. (batch number: 250101). The administration conditions are identical to those of the experimental arm in this study; however, it has no therapeutic effect.
  Other Names: A4-75mg-R
  Arms: A4-75mg-R
Drug: F-02-2-Na Tablet (150 mg) — The intervention involves the single oral administration of F-02-2-Na tablets at a dose of 150 mg, given once in a fasting state (after at least 10 hours of fasting). The drug is formulated as film-coated tablets with a strength of 50mg per tablet, manufactured by Guangdong Hengqin Novagains Biopharmaceutical Co., Ltd. (batch number: 250101). Safety and PKPD parameters will be continuously monitored for 72 hours following administration.
  Other Names: A5-150mg-T
  Arms: A5-150mg-T
Drug: F-02-2-Na Matching Placebo (150 mg) — The intervention consists of the single oral administration of a matching placebo (150 mg) for F-02-2-Na. Formulated as film-coated tablets (consistent with F-02-2-Na in appearance, color, and strength), the placebo contains no F-02-2-Na or other pharmacologically active ingredients and is manufactured by Guangdong Hengqin Novagains Biopharmaceutical Co., Ltd. (batch number: 250101). The administration conditions are identical to those of the experimental arm in this study; however, it has no therapeutic effect.
  Other Names: A5-150mg-R
  Arms: A5-150mg-R
Drug: F-02-2-Na Tablet (200 mg) — The intervention involves the single oral administration of F-02-2-Na tablets at a dose of 200 mg, given once in a fasting state (after at least 10 hours of fasting). The drug is formulated as film-coated tablets with a strength of 50mg per tablet, manufactured by Guangdong Hengqin Novagains Biopharmaceutical Co., Ltd. (batch number: 250101). Safety and PKPD parameters will be continuously monitored for 72 hours following administration.
  Other Names: A6-200mg-T
  Arms: A6-200mg-T
Drug: F-02-2-Na Matching Placebo (200 mg) — The intervention consists of the single oral administration of a matching placebo (200 mg) for F-02-2-Na. Formulated as film-coated tablets (consistent with F-02-2-Na in appearance, color, and strength), the placebo contains no F-02-2-Na or other pharmacologically active ingredients and is manufactured by Guangdong Hengqin Novagains Biopharmaceutical Co., Ltd. (batch number: 250101). The administration conditions are identical to those of the experimental arm in this study; however, it has no therapeutic effect.
  Other Names: A6-200mg-R
  Arms: A6-200mg-R
Drug: F-02-2-Na Tablet (25mg)-Multiple dose — The intervention involves the multiple oral administrations of F-02-2-Na tablets at a dose of 25mg, administered once daily for 7 consecutive days (a total of 7 administrations). The drug is formulated as film-coated tablets with a strength of 5mg/10mg per tablet, manufactured by Guangdong Hengqin Novagains Biopharmaceutical Co., Ltd. (batch number: 250101). Safety and PKPD parameters will be continuously monitored for 72 hours following administration.
  Other Names: B1-25mg-T
  Arms: B1-25mg-T
Drug: F-02-2-Na Matching Placebo (25mg) -Multiple dose — The intervention consists of the multiple oral administrations of a matching placebo (25mg) for F-02-2-Na. Formulated as film-coated tablets (consistent with F-02-2-Na in appearance, color, and strength), the placebo contains no F-02-2-Na or other pharmacologically active ingredients and is manufactured by Guangdong Hengqin Novagains Biopharmaceutical Co., Ltd. (batch number: 250101). The administration conditions are identical to those of the experimental arm in this study; however, it has no therapeutic effect.
  Other Names: B1-25mg-R
  Arms: B1-25mg-R
Drug: F-02-2-Na Tablet (50mg)-Multiple dose — The intervention involves the multiple oral administrations of F-02-2-Na tablets at a dose of 50mg, administered once daily for 7 consecutive days (a total of 7 administrations). The drug is formulated as film-coated tablets with a strength of 50mg per tablet, manufactured by Guangdong Hengqin Novagains Biopharmaceutical Co., Ltd. (batch number: 250101). Safety and PKPD parameters will be continuously monitored for 72 hours following administration.
  Other Names: B2-50mg-T
  Arms: B2-50mg-T
Drug: F-02-2-Na Matching Placebo (50mg) -Multiple dose — The intervention consists of the multiple oral administrations of a matching placebo (50mg) for F-02-2-Na. Formulated as film-coated tablets (consistent with F-02-2-Na in appearance, color, and strength), the placebo contains no F-02-2-Na or other pharmacologically active ingredients and is manufactured by Guangdong Hengqin Novagains Biopharmaceutical Co., Ltd. (batch number: 250101). The administration conditions are identical to those of the experimental arm in this study; however, it has no therapeutic effect.
  Other Names: B2-50mg-R
  Arms: B2-50mg-R
Drug: F-02-2-Na Tablet (100mg)-Multiple dose — The intervention involves the multiple oral administrations of F-02-2-Na tablets at a dose of 100mg, administered once daily for 7 consecutive days (a total of 7 administrations). The drug is formulated as film-coated tablets with a strength of 50mg per tablet, manufactured by Guangdong Hengqin Novagains Biopharmaceutical Co., Ltd. (batch number: 250101). Safety and PKPD parameters will be continuously monitored for 72 hours following administration.
  Other Names: B3-100mg-T
  Arms: B3-100mg-R
Drug: F-02-2-Na Matching Placebo (100mg) -Multiple dose — The intervention consists of the multiple oral administrations of a matching placebo (100mg) for F-02-2-Na. Formulated as film-coated tablets (consistent with F-02-2-Na in appearance, color, and strength), the placebo contains no F-02-2-Na or other pharmacologically active ingredients and is manufactured by Guangdong Hengqin Novagains Biopharmaceutical Co., Ltd. (batch number: 250101). The administration conditions are identical to those of the experimental arm in this study; however, it has no therapeutic effect.
  Other Names: B3-100mg-R
  Arms: B3-100mg-T

SUMMARY:
The primary objective of this study is to evaluate the safety, tolerability and pharmacokinetic (PK) profiles of ascending single orally administered doses of F-02-2-Na in adult subjects (to include the Mass Balance) & multiple orally administered doses of F-02-2-Na in adult subjects with Hyperuricemia.

DETAILED DESCRIPTION:
* Part 1: Approximately 39 subjects will be enrolled, 6 groups A1-A6 are predefined (A1 will enroll 3 subjects and A2&A6 will enroll 6 subjects, A3A4A5 will enroll 8 subjects). The planned dose escalation of F-02-2-Na will include 6-ascending single-dose cohorts with tentative PO doses ranging from 0.5 mg to 200 mg. Subjects in each SAD cohort will be randomly assigned to receive active drug or matching placebo in a 2:1 or 3:1 ratio (n=2 or 4 or 6 subjects to receive F-02-2-Na, n=1 or 2 subjects will be administered placebo).Safety and PKPD assessments will continue for 72 hours post dose, with discharge from the Phase I Clinical Research Center following completion of all 72-hour procedures on Day 4. Subjects will receive a phone call for an End-of-Study (EOS) follow-up on Day 7 (±1 day).In SAD A3 (25 mg), collected blood, urine, and feces will be used for the mass balance study.
* Part 2: Approximately 30 subjects will be enrolled.Three dose groups (B1~B3) are predefined, with 10 subjects per group (including 2 subjects receiving placebo). The administration doses are 25 mg, 50 mg, and 100 mg respectively, administered once daily for 7 consecutive days (a total of 7 administrations).After subjects complete the collection of pharmacokinetic and pharmacokinetics blood & urine samples at 72.0 hours post-administration and undergo relevant examinations, they may leave the Phase I Clinical Research Center upon completion of all tests .

ELIGIBILITY:
Inclusion Criteria:

* For Healthy Adult Subjects
* 1.The subjects should fully understand the purpose, nature, process of the study and the possible adverse reactions, voluntarily act as subjects, and sign the informed consent form before the start of any research procedures.
* 2.Healthy male or female subjects aged 18 to 45 years old (inclusive).
* 3.The body weight for male and female subjects should be ≥ 50.0 kg and ≥ 45.0 kg, respectively; the body mass index (BMI) should be between 19 kg/m² and 26 kg/m² (inclusive).
* 4.The subjects should have normal results or abnormal results without clinical significance in vital signs check, physical examination, clinical laboratory tests (Complete Blood Count(CBC), urine analysis, blood biochemistry, coagulation panel, free thyroid function tests), chest X-ray, liver and renal color ultrasound and 12-lead electrocardiogram.
* 5. Normal renal function as determined by Investigator following review of clinical laboratory test results, including eGFR ≥ 90 mL/min/1.73 m².
* 6. The subjects (including male subjects) should have no plans for having children from screening until 6 months after the last dose and should voluntarily take effective contraceptive measures and have no plans for sperm or egg donation.
* 7. The subjects should be able to communicate well with the researchers and understand and comply with the requirements of this study.
* For Adult Subjects with Hyperuricemia
* 1. The subjects should fully understand the purpose, nature, process of the study and the possible adverse reactions, voluntarily act as subjects, and sign the informed consent form before the start of any research procedures.
* 2. Male or female subjects aged 18 to 45 years (inclusive).
* 3. Body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females; Body Mass Index (BMI) between 18 kg/m² and 28 kg/m² (inclusive).
* 4. Subjects with results from vital signs check, physical examination, clinical laboratory tests (except for serum uric acid), chest X-ray, liver ultrasonography, renal ultrasonography, and 12-lead electrocardiogram that show no abnormalities or only abnormalities of no clinical significance.
* 5. Estimated Glomerular Filtration Rate (eGFR) > 90 mL/min/1.73m² (calculated using the CKD-EPI Creatinine Equation).
* 6. The subjects (including male subjects) should have no plans for having children from screening until 6 months after the last dose and should voluntarily take effective contraceptive measures and have no plans for sperm or ova donation.
* 7. Does not meet the 2015 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) Gout Classification Criteria; however, two fasting serum uric acid levels during the screening period are both ≥ 540 μmol/L (as determined by the study center's test results), and the investigator deems the subject in need of long-term uric acid-lowering therapy.

Exclusion Criteria:

* 1. Subjects with a specific allergic history (such as asthma, urticaria, eczema, etc.) or those with an allergic constitution (such as those known to be allergic to two or more substances), or those with a known history of allergy to F-02-2-Na and related excipients (ascertained through inquiry).
* 2. Subjects who have had an acute illness within two weeks before the first drug administration (ascertained through inquiry).
* 3. Subjects with diseases of important organs or systems (including but not limited to liver, kidney, nervous system, blood, endocrine system, lungs, immune system, mental health, cardiovascular and cerebrovascular system, gastrointestinal tract, skin, metabolism, bone and joints, etc.) that are considered clinically significant by the researcher, or those with a history of such serious diseases; or those with a history of tumor (ascertained through inquiry).
* 4. Subjects with a history of gastrointestinal, liver, kidney, and thyroid diseases that can affect drug absorption or metabolism (ascertained through inquiry).
* 5. Subjects with a history of gout (ascertained through inquiry).
* 6. Subjects who have used any medications (including any prescription drugs, over-the-counter drugs, traditional Chinese herbal medicines) and health products within two weeks before the first drug administration (ascertained through inquiry).
* 7. Subjects who have used any mercaptopurine hydrate or thiopurine drugs within four weeks before the study (ascertained through inquiry).
* 8. Subjects who have heavily consumed, within 2 weeks prior to the first dose, or ingested within 48 hours prior to dosing, beverages containing caffeine or alcohol, or foods known to affect drug metabolism (such as chocolate, pitaya, mango, pomelo, carambola, guava, orange, grapefruit, or grapefruit products).(ascertained through inquiry)
* 9. Subjects who have undergone major surgical procedures (excluding diagnostic surgical procedures) within six months before the study , or those who plan to have surgery during the research period, or those who have undergone surgeries that, in the judgment of the researcher, can affect drug absorption, distribution, metabolism, and excretion (ascertained through inquiry).
* 10. Subjects who have received vaccination within three months before the study (ascertained through inquiry).
* 11. Subjects who have participated in any other clinical trial within 3 months prior to the current study. (Note: The end date is defined as the date of completion/exit from the previous clinical trial.) (ascertained through inquiry).
* 12. Subjects who have donated blood within three months before the study, or those whose total blood loss due to blood donation or other reasons has reached or exceeded 400 mL within six months (ascertained through inquiry).
* 13. Subjects who, on average, consumed more than 14 units of alcohol per week over the past year, or those unable to abstain from alcohol during the study period, or individuals with a breath alcohol test result greater than 0.0 mg/100 mL (ascertained through inquiry/examination).
* 14. Subjects who smoke more than 5 cigarettes per day on average within three months before the study, or those who cannot stop using any tobacco products during the study (ascertained through inquiry).
* 15. Subjects with a history of drug abuse (including the repeated and excessive use of various narcotic drugs and psychotropic substances for non-medical purposes) or positive results in drug abuse screening (including morphine, methamphetamine, ketamine, MDMA (3,4-methylenedioxymethamphetamine), cannabis (tetrahydrocannabinolic acid), etc.) within the past year (ascertained through inquiry and examination).
* 16. Subjects with a positive result in any item of the infectious disease examination during the screening period (including hepatitis B surface antigen, hepatitis C antibody, human immunodeficiency virus antibody, and treponema pallidum antibody) (examination).
* 17. Subjects who cannot tolerate venipuncture/indwelling needle or those with a history of fainting at the sight of needles or blood (ascertained through inquiry).
* 18. Subjects with difficult venous blood collection (ascertained through inquiry).
* 19. Subjects with lactose intolerance (ascertained through inquiry). 20. Subjects with special dietary requirements and who cannot accept the unified diet (ascertained through inquiry).
* 21. Subjects with dysphagia (ascertained through inquiry).
* 22. Other subjects are deemed unsuitable for participation by the researcher.
* 23. In addition to the above requirements, female subjects who meet the following conditions should also be excluded:
* a. Those who have used oral contraceptives within 30 days before the study ( ascertained through inquiry ) .
* b. Those who have used long-acting estrogen or progesterone injections ( including progesterone-containing intrauterine contraceptive devices ) or implanted tablets within 6 months before the study (ascertained through inquiry ) .
* c. Those who have unprotected sexual intercourse with their partners within 14 days before the study ( ascertained through inquiry ) .
* d. Those with a positive blood pregnancy test result ( examination ) .
* e. Pregnant or lactating women ( ascertained through inquiry ) .

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability: Adverse Events (AEs) of ascending single and multiple oral doses of F-02-2-Na in adult subjects. | 0-72 hours post dose
  Incidence, severity, and seriousness of adverse events (AEs) following ascending single and multiple oral doses of F-02-2-Na in adult subjects.
Safety and Tolerability: Concomitant Medications of ascending single and multiple oral doses in Adult Subjects | 0-72 hours post dose
  Proportion of adult Subjects Using Concomitant Medications During Treatment during treatment with ascending single and multiple oral doses of F-02-2-Na.
Safety and Tolerability: Electrocardiogram (ECG) Findings ascending single and multiple oral doses of F-02-2-Na in Adult Subjects | From pre-dose (baseline) to 72 hours after the last dose.
  Proportion of adult subjects with abnormal findings in electrocardiogram (ECG) parameters (including PR interval, QRS duration, QT/QTc interval, heart rate, and rhythm) following ascending single and multiple oral doses of F-02-2-Na.
Proportion of subjects with abnormal hematology findings following ascending single and multiple oral doses of F-02-2-Na. | From pre-dose (baseline) to 72 hours after the last dose.
  Proportion of subjects with clinically significant abnormalities in hematology parameters (e.g., hemoglobin, hematocrit, red blood cell count, white blood cell count with differential, platelet count).
Proportion of subjects with abnormal coagulation findings following ascending single and multiple oral doses of F-02-2-Na. | From pre-dose (baseline) to 72 hours after the last dose.
  Proportion of adult subjects with clinically significant abnormalities in coagulation parameters (e.g., PT, INR, aPTT).
Proportion of subjects with abnormal urinalysis findings following ascending single and multiple oral doses of F-02-2-Na. | From pre-dose (baseline) to 72 hours after the last dose.
  Proportion of adult subjects with clinically significant abnormalities in urinalysis parameters (e.g., protein, glucose, blood, microscopic examination)
Proportion of subjects with abnormal clinical chemistry findings following ascending single and multiple oral doses of F-02-2-Na | pre-dose (baseline) to 72 hours after the last dose
  Incidence of clinically significant abnormalities in clinical chemistry parameters (e.g., sodium, potassium, chloride, calcium, ALT, AST, total bilirubin, alkaline phosphatase, creatinine, BUN, glucose).
Proportion of subjects with abnormal renal morphology following administration of F-02-2-Na | From pre-dose (baseline) to 72 hours after the last dose
  Proportion of adult subjects with abnormal renal morphology as assessed by Renal Color Doppler Ultrasonography (Renal CDU) following ascending single and multiple oral doses of F-02-2-Na
Proportion of subjects with abnormal pelvicalyceal system findings following administration of F-02-2-Na | From pre-dose (baseline) to 72 hours post dose
  Proportion of adult subjects with abnormal pelvicalyceal system findings as assessed by Renal CDU following ascending single and multiple oral doses of F-02-2-Na.
Proportion of subjects with abnormal renal vascular hemodynamics following administration of F-02-2-Na | From pre-dose (baseline) to 72 hours post dose
  Proportion of adult subjects with abnormal renal vascular hemodynamics as assessed by Renal CDU following ascending single and multiple oral doses of F-02-2-Na.
Pharmacokinetic Profile: Maximum Plasma Concentration (Cmax) of F-02-2-Na in healthy Adult Subjects | From pre-dose (baseline) to 72 hours post dose
  To evaluate the Pharmacokinetic parameters:Maximum plasma concentration (Cmax) of F-02-2-Na following ascending single oral doses in healthy adult subjects.
Area Under the Concentration (AUC0-t) of F-02-2-Na in healthy Adult Subjects | From pre-dose (baseline) to 72 hours post dose
  To evaluate the Pharmacokinetic parameters:Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (AUC0-t) of F-02-2-Na following ascending single oral doses in healthy adult subjects.
Pharmacokinetic Profile: Area Under the Concentration (AUC0-∞) of F-02-2-Na in healthy Adult Subjects | From pre-dose (baseline) to 72 hours post dose
  To evaluate the Pharmacokinetic parameters: Area Under the Concentration-Time Curve from Time 0 to Extrapolated Infinity (AUC0-∞) of F-02-2-Na following ascending single oral doses in healthy adult subjects.
Pharmacokinetic Profile: Time to Maximum Plasma Concentration (Tmax) of F-02-2-Na in Adult Subjects | From pre-dose (baseline) to 72 hours after the last dose
  To evaluate the Pharmacokinetic parameters:Time to reach maximum plasma concentration (Tmax) of F-02-2-Na following ascending single and multiple oral doses in adult subjects.
Pharmacokinetic Profile: Terminal Elimination Half-Life (t1/2) of F-02-2-Na in Adult Subjects | From pre-dose (baseline) to 72 hours after the last dose
  To evaluate the Pharmacokinetic Parameters:Terminal elimination half-life (t1/2) of F-02-2-Na following ascending single and multiple oral doses in adult subjects.
Pharmacokinetic Profile: Mean Residence Time from Time 0 to Last Quantifiable Concentration (MRT0-t) of F-02-2-Na in Healthy Adult Subjects | From pre-dose (baseline) to 72 hours post dose.
  To evaluate the pharmacokinetic parameters:Mean residence time from time 0 to the last quantifiable concentration (MRT0-t) of F-02-2-Na following ascending single oral doses in healthy adult subjects.
Pharmacokinetic Profile: Mean Residence Time from Time 0 to Extrapolated Infinity (MRT0-∞) of F-02-2-Na in Adult Subjects | From pre-dose (baseline) to 72 hours post dose
  To evaluate the pharmacokinetic parameters: Mean residence time from time 0 to extrapolated infinity (MRT0-∞) of F-02-2-Na following ascending single and multiple oral doses in adult subjects.
Pharmacokinetic Profile: Apparent Clearance/Bioavailability (CL/F) of F-02-2-Na in Adult Subjects | From pre-dose (baseline) to 72 hours after the last dose
  To evaluate the pharmacokinetic parameters: Apparent clearance normalized to bioavailability (CL/F) of F-02-2-Na following ascending single and multiple oral doses in adult subjects.
Pharmacokinetic Profile: Apparent Volume of Distribution at Steady State (Vz/F) of F-02-2-Na in Adult Subjects | From pre-dose (baseline) to 72 hours after the last dose
  To evaluate the pharmacokinetic parameters: Apparent volume of distribution at steady state (Vz/F) of F-02-2-Na following ascending single and multiple oral doses in adult subjects.
Pharmacokinetic Profile: Terminal Elimination Rate Constant (Kel) of F-02-2-Na in Healthy Adult Subjects | From pre-dose (baseline) to 72 hours after the last dose
  To evaluate the pharmacokinetic parameters: Terminal elimination rate constant (Kel) of F-02-2-Na following ascending single oral doses in healthy adult subjects.
Pharmacokinetic Profile: Minimum Steady-State Plasma Concentration (Css_min) of F-02-2-Na in Adult Subjects with Hyperuricemia | From pre-dose (baseline) to 72 hours after the last dose
  To evaluate the pharmacokinetic parameters: Minimum Steady-State Plasma Concentration (Css_min) of F-02-2-Na following ascending multiple oral doses in Adult Subjects with Hyperuricemia.
Pharmacokinetic Profile: Maximum Steady-State Plasma Concentration (Css_max) of F-02-2-Na in Adult Subjects with Hyperuricemia | From pre-dose (baseline) to 72 hours after the last dose.
  To evaluate the pharmacokinetic parameters: Maximum Steady-State Plasma Concentration (Css_max) of F-02-2-Na following ascending multiple oral doses in Adult Subjects with Hyperuricemia.
Pharmacokinetic Profile: Average Steady-State Plasma Concentration (Css_av) of F-02-2-Na in Adult Subjects with Hyperuricemia | From pre-dose (baseline) to 72 hours after the last dose.
  To evaluate the pharmacokinetic parameters: Average Steady-State Plasma Concentration (Css_av) of F-02-2-Na following ascending multiple oral doses in Adult Subjects with Hyperuricemia.
Pharmacokinetic Profile: Area Under the Concentration (AUCss,0-t) of F-02-2-Na in Adult Subjects with Hyperuricemia | From pre-dose (baseline) to 72 hours after the last dose
  To evaluate the pharmacokinetic parameters: Area Under the Steady-State Concentration-Time Curve from Time 0 to Last Quantifiable Concentration (AUCss,0-t) of F-02-2-Na following ascending multiple oral doses in Adult Subjects with Hyperuricemia.
Pharmacokinetic Profile: Area Under the Concentration (AUCss,0-∞) of F-02-2-Na in Adult Subjects with Hyperuricemia | From pre-dose (baseline) to 72 hours after the last dose
  To evaluate the pharmacokinetic parameters: Area Under the Steady-State Concentration-Time Curve from Time 0 to Extrapolated Infinity(AUCss,0-∞) of F-02-2-Na following ascending multiple oral doses in Adult Subjects with Hyperuricemia.
Pharmacokinetic Profile: Area Under the Concentration (AUC0-tau) of F-02-2-Na in Adult Subjects with Hyperuricemia | From pre-dose (baseline) to 72 hours after the last dose
  To evaluate the pharmacokinetic parameters: Area Under the Concentration-Time Curve over One Dosing Interval (AUC0-tau) of F-02-2-Na following ascending multiple oral doses in Adult Subjects with Hyperuricemia.
Pharmacokinetic Profile: Accumulation Ratio (Rac) of F-02-2-Na in Adult Subjects with Hyperuricemia | From pre-dose (baseline) to 72 hours after the last dose
  To evaluate the pharmacokinetic parameters: Accumulation Ratio (Rac) of F-02-2-Na following ascending multiple oral doses in Adult Subjects with Hyperuricemia.
Pharmacokinetic Profile: Degree of Fluctuation (DF) of F-02-2-Na in Adult Subjects with Hyperuricemia | From pre-dose (baseline) to 72 hours after the last dose
  To evaluate the pharmacokinetic parameters: Degree of Fluctuation (DF) of F-02-2-Na following ascending multiple oral doses in Adult Subjects with Hyperuricemia.

SECONDARY OUTCOMES:
Mass Balance: Total Renal Excretion Amount of F-02-2-Na in Healthy Adult Subjects | From pre-dose (baseline) to 72 hours post dose.
  Total amount of F-02-2-Na excreted via the renal route (expressed as absolute amount or percentage of administered dose), estimated from urinary drug concentrations in healthy adult subjects.
Mass Balance: Fecal Excretion Rate of F-02-2-Na in Healthy Adult Subjects | From pre-dose (baseline) to 72 hours post dose.
  Rate of F-02-2-Na excretion via the fecal route, estimated from fecal drug concentrations in healthy adult subjects.
Mass Balance: Total Fecal Excretion Amount of F-02-2-Na in Healthy Adult Subjects | From pre-dose (baseline) to 72 hours post dose.
  Total amount of F-02-2-Na excreted via the fecal route (expressed as absolute amount or percentage of administered dose), estimated from fecal drug concentrations in healthy adult subjects.
Explore the dose-exposure-effect relationship：Correlation between Exposure Parameters of F-02-2-Na and Serum Uric Acid (sUA) Reduction in Adult Subjects | From pre-dose (baseline) to 72 hours after the last dose.
  Correlation analysis between pharmacokinetic exposure parameters (e.g., Cmax, AUC0-∞, AUCss,0-tau) of F-02-2-Na tablets and the degree of serum uric acid (sUA) reduction in adult subjects. The correlation will be evaluated using statistical methods.
Exploration of Potential Biomarkers Associated with the Pharmacodynamics of F-02-2-Na in Adult Subjects | From pre-dose (baseline) to 72 hours after the last dose.
  Exploration and identification of potential biomarkers (e.g., molecular, genetic, or biochemical markers) associated with the pharmacodynamic effects of F-02-2-Na tablets in adult subjects, through analysis of biological samples (e.g., blood, urine) collected during the study.
Absolute Change in Serum Uric Acid (sUA) Levels in Adult Subjects After Single and Multiple Oral Administrations of F-02-2-Na | From pre-dose (baseline) to 72 hours after the last dose.
  To evaluate the absolute change in serum uric acid (sUA) levels in adult subjects after single and multiple oral administrations of F-02-2-Na. The absolute change is calculated as the difference between sUA levels at each predefined time point and the baseline sUA level (absolute change = sUA level at predefined time point - baseline sUA level).
Percentage Change in Serum Uric Acid (sUA) Levels in Adult Subjects After Single and Multiple Oral Administrations of F-02-2-Na | From pre-dose (baseline) to 72 hours after the last dose.
  To evaluate the percentage change in serum uric acid (sUA) levels in adult subjects after single and multiple oral administrations of F-02-2-Na. The percentage change is calculated relative to the baseline sUA level at each predefined time point (percentage change = [(sUA level at predefined time point - baseline sUA level)/baseline sUA level] × 100%).
Uric Acid Excretion (AeUR) in Adult Subjects After Single and Multiple Oral Administrations of F-02-2-Na | From pre-dose (baseline) to 72 hours after the last dose.
  To evaluate the uric acid excretion (AeUR) in adult subjects after single and multiple oral administrations of F-02-2-Na. AeUR is defined as the total amount of uric acid excreted in urine within a specified time period (e.g., 24 hours or predefined intervals after administration), reflecting the cumulative excretion capacity of uric acid.
Uric Acid Clearance Rate (CLUR) in Adult Subjects After Single and Multiple Oral Administrations of F-02-2-Na | From pre-dose (baseline) to 72 hours after the last dose.
  To evaluate the uric acid clearance rate (CLUR) in adult subjects after single and multiple oral administrations of F-02-2-Na. CLUR is calculated as the ratio of uric acid excretion rate to serum uric acid concentration (CLUR = AeUR / AUC_sUA), reflecting the efficiency of renal uric acid clearance, with the unit of volume per unit time (e.g., mL/min).
Area Under the Curve (AUC) of Serum Uric Acid (sUA) Dynamic Change Curve in Adult Subjects After Single and Multiple Oral Administrations of F-02-2-Na | From pre-dose (baseline) to 72 hours after the last dose.
  To evaluate the area under the curve (AUC) of the serum uric acid (sUA) dynamic change curve in adult subjects after single and multiple oral administrations of F-02-2-Na. AUC is calculated by integrating the sUA concentration-time curve over a predefined time period (e.g., AUC₀-t, AUC₀-∞), reflecting the total exposure level of sUA during the observation period, with the unit of concentration × time (e.g., μmol·h/L).
Total 24-Hour Uric Acid Excretion in Adult Subjects After Single and Multiple Oral Administrations of F-02-2-Na | From pre-dose (baseline) to 72 hours after the last dose.
  To evaluate the total 24-hour uric acid excretion in adult subjects after single and multiple oral administrations of F-02-2-Na. It is determined by collecting 24-hour urine samples, measuring the uric acid concentration in the urine, and calculating the total amount of uric acid excreted in 24 hours (Total 24-hour uric acid excretion = Urine uric acid concentration × 24-hour urine volume), with the unit of mass (e.g., mg/24h or mmol/24h).

CONTACTS AND LOCATIONS:
Overall Officials: Junyan Wu, MS, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Donghui Zheng, MM, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
This is a Phase I exploratory study, and the data involves core information related to drug development. Therefore, there are no current plans to share Individual Participant Data (IPD).

REFERENCES:
- [Background] Lee HA, Yu KS, Park SI, Yoon S, Onohara M, Ahn Y, Lee H. URC102, a potent and selective inhibitor of hURAT1, reduced serum uric acid in healthy volunteers. Rheumatology (Oxford). 2019 Nov 1;58(11):1976-1984. doi: 10.1093/rheumatology/kez140. PMID 31056705
- [Background] Hall J, Gillen M, Yang X, Shen Z. Pharmacokinetics, Pharmacodynamics, and Tolerability of Concomitant Administration of Verinurad and Febuxostat in Healthy Male Volunteers. Clin Pharmacol Drug Dev. 2019 Feb;8(2):179-187. doi: 10.1002/cpdd.463. Epub 2018 Apr 24. PMID 29688628
- [Background] Ding R, Chen L, Li X, Xiong T, Chen H, Hu X, Li Y, Zhou Y, Liu K, Wu J, Jiang F, Peng Q. A Phase I Study to Evaluate the Pharmacokinetic Drug-Drug Interaction of HP501, Febuxostat, and Colchicine in Male Chinese Patients with Hyperuricemia. Clin Drug Investig. 2023 Jun;43(6):401-411. doi: 10.1007/s40261-023-01274-7. Epub 2023 May 30. PMID 37248357
- [Background] Wang Z, Li X, Jin Y, Liu R, Di X, Zhou Y, Wang Y, Fan L, Chen Y, Wang Y, Zheng L. Safety, Efficacy, and Pharmacokinetics of HP501 in Healthy Volunteers and Hyperuricemic Patients: A Phase I/IIa Study. J Clin Endocrinol Metab. 2022 May 17;107(6):1667-1678. doi: 10.1210/clinem/dgac032. PMID 35106590